CLINICAL TRIAL: NCT07194746
Title: The Prevalence of Neck and Low Back Pain in Staff of the Faculty of Medical Sciences Teaching & Research Complex at the University of the West Indies Mona Campus
Brief Title: The Prevalence of Neck and Low Back Pain in FMSTRC Staff At the UWI Mona
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Collaborators: The University of The West Indies, Mona (Unknown)
Responsible Party: Principal Investigator, Paula Dawson, MBBS, Head, Physical Medicine and Rehabilitation. Principal Investigator, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Neck Pain; Back Pain; Musculoskeletal Pain; Low Back Pain; Spine; Work Related Illnesses; Work Related Musculoskeletal Disorders
Keywords: neck pain; back pain; Musculoskeletal pain; low back pain; spinal health; work related musculoskeletal disorders
MeSH Terms: conditions — Neck Pain; Back Pain; Musculoskeletal Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Control (Group A) (Experimental): All participants will complete the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) to assess the frequency, discomfort and interference with work due to musculoskeletal pain; the Numeric Rating Scale (NRS) to assess for perceived pain; as well as Questionnaire A to assess their knowledge, attitude and practice towards musculoskeletal problems of neck or low back pain. Participants who are found to have neck or low back pain will be randomised into two (2) groups: a clinical control group (Group A) and an intervention group (Group B). Group A will be given a non-specific spine exercise program over an eight (8) week period after which time, participants will be reassessed using the CMDQ and NRS, as well as a Questionnaire B to evaluate for changes in their knowledge, attitude and practice towards musculoskeletal problems of the neck and low back pain.
  Interventions: Behavioral: Clinical Control Group (Group A)
- Spine Exercise Program (Group B) (Experimental): All participants will complete the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) to assess the frequency, discomfort and interference with work due to musculoskeletal pain; the Numeric Rating Scale (NRS) to assess for perceived pain; as well as Questionnaire A to assess their knowledge, attitude and practice towards musculoskeletal problems of neck or low back pain. Participants who are found to have neck or low back pain will be randomised into two (2) groups: a clinical control group (Group A) and an intervention group (Group B). Group B will be given a standardised spine-specific exercise program over an eight (8) week period, after which time they will be be reassessed using the CMDQ and NRS, as well as Questionnaire B to evaluate for changes in their knowledge, attitude and practice towards musculoskeletal problems of the neck and low back pain, having received the intervention.
  Interventions: Behavioral: Spine Exercise Program (Group B)

INTERVENTIONS:
Behavioral: Clinical Control Group (Group A) — The participants who reported the presence of neck or low back pain and were assigned to the clinical control group (Group A) after randomisation will receive a non-specific spine exercise program provided in a handout. The interventional group (Group B) will be asked to keep the standardised spine-specific exercise program confidential and not share with the control group (Group A). After eight (8) weeks, Group A participants will receive: the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) to assess for changes in the frequency, discomfort and interference with work due to musculoskeletal pain; a Questionnaire B, to ascertain any changes in their pain level using the Numeric Rating Scale (NRS); as well as their knowledge, attitude and practice towards musculoskeletal problems of the neck and low back pain.
  Arms: Clinical Control (Group A)
Behavioral: Spine Exercise Program (Group B) — The standardised spine-specific exercise program will be provided in a handout and given only to the intervention group (Group B), and will include specific spine basic neck or low back exercises to be done three (3) times per week, as well as brief stretching exercises, to be done during periods of sitting for greater than sixty (60) minutes. The selected participants will be asked to comply with instructions on the handout. Participants who experience worsening of their symptoms, or who develop new symptoms will be assessed as having an adverse outcome and will be withdrawn from the study and referred for evaluation and treatment if necessary.
  Arms: Spine Exercise Program (Group B)

SUMMARY:
The purpose of this study is to identify the prevalence of neck and low back pain in full-time staff in the Faculty of Medical Sciences Teaching and Research Complex at The University of the West Indies, Mona; to assess their knowledge, attitude and practice of good spine health and to determine the outcome of a standardised spine exercise program on staff experiencing neck and low back pain, using a prospective randomised control design.

DETAILED DESCRIPTION:
Musculoskeletal pain is a widespread problem in varied occupational groups. Globally, low back pain is among the leading causes of disability and morbidity in adults, contributing to a significant health care and socioeconomic burden. It is strongly associated with lost workdays, reduced productivity, and increased workers' compensation claims (Samad NIA AH, 2010) (GA, 2005). Studies suggest that approximately 37% of low back pain cases are occupation related, and the lifetime prevalence of neck pain is estimated to be as high as 70%. Occupational risk factors vary across work groups(Cagnie B DL, 2007). Office and academic staff are prone to neck pain due to prolonged sitting, forward head posture, and sustained computer use. Ancillary workers, such as cleaners and those performing manual tasks, are more often affected by low back pain linked to repetitive lifting, awkward postures, and whole-body vibration. For example, Chang (2012) reported that nearly 90% of cleaners experienced musculoskeletal discomfort, with 37.8% citing low back pain as their main complaint. Lifestyle and environmental factors also contribute. Green (2016) found a strong association between smoking and back pain: prevalence was 23.5% in never-smokers, 33.1% in former smokers, and 36.9% in current smokers. Genetic influences are also significant, with Lier (2015) showing that parental spinal pain was consistently linked to higher risk of chronic pain in adult offspring. Evidence supports targeted interventions. Sihawong et al. (2014) demonstrated that office workers who participated in a structured stretching and endurance program had a reduced incidence of low back pain. Similarly, a randomised controlled trial by Shariat (2018) found significant reductions in both neck and back pain scores among office workers following a combined program of stretching and ergonomic modifications. Despite this growing body of evidence, there is a lack of published research from Jamaica and the wider Caribbean on the prevalence of neck and low back pain among university staff. These conditions not only impair physical health but can also affect social and occupational functioning, leading to decreased quality of life. This study seeks to determine the prevalence of neck and low back pain among full-time staff in the Faculty of Medical Sciences Teaching and Research Complex at The University of the West Indies,Mona. It also aims to assess knowledge, attitudes, and practices regarding spine health, and to evaluate the effects of a standardised spine-specific exercise program on musculoskeletal discomfort. A prospective randomised controlled trial will be conducted with staff who report neck and low back pain. Participants will be randomised into a control group (Group A), which will receive a non-specific spine exercise program, or an intervention group (Group B), which will complete an eight (8) weeks standardised spine-specific exercise program. The non-specific spine exercise program will aid in minimising the placebo effect. This program focuses on stretching, flexibility, and core strengthening exercises to improve posture, spinal stability, and functional capacity. Data will be collected using Questionnaires A and B, the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ), and the Numeric Rating Scale (NRS). Outcomes between groups will then be compared to determine the effectiveness of the specific spine exercise program in reducing discomfort and improving spine health practices among the participants. Confidentiality will be strictly observed. Each participant will be assigned a study number, and only demographic, clinical, and outcome data will be recorded. All data will be securely stored on REDCap, a password-protected, web-based platform that complies with national data protection standards. Statistical analysis will be conducted using SPSS, and all records will be securely destroyed three years after study completion.

ELIGIBILITY:
Inclusion Criteria

1. All full time academic/office/supplementary/ancillary staff employed to the Faculty of Medical Science, Training and Research Complex, UWI, Mona.
2. Individuals with a willingness to adhere to exercise program given in a handout.
3. Individuals age 18-65
4. Individuals with at least 1 year experience in their current position.

Exclusion Criteria

1. Individuals with a history of having spine surgery
2. Individuals previously diagnosed with a spine pathology
3. Individuals currently receiving physiotherapy for a spine problem

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender men and cisgender women
Enrollment: 200 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) | From enrollment to the end of treatment at eight (8) weeks
  The Cornell Musculoskeletal Discomfort Questionnaire measures the frequency, discomfort and interference with work due to musculoskeletal pain, as reported by participants. The individually reported frequency score is then multiplied by the discomfort score and by the interference score to determine overall severity of pain experienced. This tallied score is then classified by severity into: no discomfort (0), mild (1 to 4.5), moderate (5 to 14), severe (15 - 45) and very severe (45 or higher). All participants will complete this assessment upon enrollment, as well as after an eight (8) week period of treatment, to evaluate any changes in their reported scores.

SECONDARY OUTCOMES:
Knowledge, Attitude and Practice towards Musculoskeletal Problems of Neck and Low back Pain (Questionnaire A) | Done at the time of enrollment (Baseline)
  Questionnaire A is a self-administered general questionnaire used to evaluate knowledge, attitude and practice towards musculoskeletal problems of neck and low back pain.
Change from Baseline in Knowledge, Attitude and Practice Towards Musculoskeletal Problems of Neck and Low Back Pain (Questionnaire B) | From Enrollment to the end of treatment at 8 weeks
  Questionnaire B is a self-administered general questionnaire used to evaluate changes in knowledge, attitude and practice towards musculoskeletal problems of neck and low back pain.
Change from Baseline in the Numeric Rating Scale (NRS) | From Enrollment to the end of treatment at 8 weeks
  The Numeric Rating Scale is a reliable and valid, unidimensional 11-point scale used for patient self-reporting of perceived pain. Its scale uses integers which range from zero (0) to ten (10), where 0 represents no pain, and 10 represents the worst imaginable pain. This is then categorised into mild (1-3), moderate (4-6), and severe (7-10). All participants will complete this assessment upon enrollment, as well as after an eight (8) week period of treatment, to evaluate any changes in their perceived pain. This scale is from public domains and as such, permission for its use is not required.

CONTACTS AND LOCATIONS:
Overall Officials: Paula U. A. Dawson, MBBS, Diplomate ABPMR, Principal Investigator — Division of Physical Medicine and Rehabilitation, Faculty of Medical Sciences, The University of the West Indies, Mona, Jamaica.
Locations (1):
- Faculty of Medical Sciences Teaching and Research Complex, University of The West Indies-Mona Campus, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007 Oct 2;147(7):478-91. doi: 10.7326/0003-4819-147-7-200710020-00006. PMID 17909209
- [Background] Shariat A, Cleland JA, Danaee M, Kargarfard M, Sangelaji B, Tamrin SBM. Effects of stretching exercise training and ergonomic modifications on musculoskeletal discomforts of office workers: a randomized controlled trial. Braz J Phys Ther. 2018 Mar-Apr;22(2):144-153. doi: 10.1016/j.bjpt.2017.09.003. Epub 2017 Sep 6. PMID 28939263
- [Background] Lier R, Nilsen TI, Vasseljen O, Mork PJ. Neck/upper back and low back pain in parents and their adult offspring: Family linkage data from the Norwegian HUNT Study. Eur J Pain. 2015 Jul;19(6):762-71. doi: 10.1002/ejp.599. Epub 2014 Sep 29. PMID 25263611
- [Background] Green BN, Johnson CD, Snodgrass J, Smith M, Dunn AS. Association Between Smoking and Back Pain in a Cross-Section of Adult Americans. Cureus. 2016 Sep 26;8(9):e806. doi: 10.7759/cureus.806. PMID 27790393
- [Background] Chang JH, Wu JD, Liu CY, Hsu DJ. Prevalence of musculoskeletal disorders and ergonomic assessments of cleaners. Am J Ind Med. 2012 Jul;55(7):593-604. doi: 10.1002/ajim.22064. Epub 2012 Apr 27. PMID 22544565
- [Background] Naing L, Nordin RB, Abdul Rahman H, Naing YT. Sample size calculation for prevalence studies using Scalex and ScalaR calculators. BMC Med Res Methodol. 2022 Jul 30;22(1):209. doi: 10.1186/s12874-022-01694-7. PMID 35907796
- [Background] Gordon R, Bloxham S. A Systematic Review of the Effects of Exercise and Physical Activity on Non-Specific Chronic Low Back Pain. Healthcare (Basel). 2016 Apr 25;4(2):22. doi: 10.3390/healthcare4020022. PMID 27417610
- [Background] Herman Miller Research Corporation. (1989). How office workers spend their time and position themselves. Internal document.
- [Background] Erdinc O HK, Ozkaya M. CROSS-CULTURAL ADAPTATION,VALIDITY AND RELIABILITY OFCORNELL MUSCULOSKELETAL DISCOMFORT QUESTIONNAIRE (CMDQ) IN TURKISH LANGUAGE. 2008.
- [Background] Ariens GA, van Mechelen W, Bongers PM, Bouter LM, van der Wal G. Physical risk factors for neck pain. Scand J Work Environ Health. 2000 Feb;26(1):7-19. doi: 10.5271/sjweh.504. PMID 10744172
- [Background] Lis AM, Black KM, Korn H, Nordin M. Association between sitting and occupational LBP. Eur Spine J. 2007 Feb;16(2):283-98. doi: 10.1007/s00586-006-0143-7. Epub 2006 May 31. PMID 16736200
- [Background] Lorusso A, Vimercati L, L'abbate N. Musculoskeletal complaints among Italian X-ray technology students: a cross-sectional questionnaire survey. BMC Res Notes. 2010 Apr 24;3:114. doi: 10.1186/1756-0500-3-114. PMID 20416101
- [Background] Smith DR, Wei N, Ishitake T, Wang RS. Musculoskeletal disorders among Chinese medical students. Kurume Med J. 2005;52(4):139-46. doi: 10.2739/kurumemedj.52.139. PMID 16639985
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Nonpharmacologic therapies for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):492-504. doi: 10.7326/0003-4819-147-7-200710020-00007. PMID 17909210
- [Background] O'Sullivan PB, Phyty GD, Twomey LT, Allison GT. Evaluation of specific stabilizing exercise in the treatment of chronic low back pain with radiologic diagnosis of spondylolysis or spondylolisthesis. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2959-67. doi: 10.1097/00007632-199712150-00020. PMID 9431633
- [Background] Chiu TT, Ku WY, Lee MH, Sum WK, Wan MP, Wong CY, Yuen CK. A study on the prevalence of and risk factors for neck pain among university academic staff in Hong Kong. J Occup Rehabil. 2002 Jun;12(2):77-91. doi: 10.1023/a:1015008513575. PMID 12014228
- [Background] Sihawong R, Janwantanakul P, Jiamjarasrangsi W. A prospective, cluster-randomized controlled trial of exercise program to prevent low back pain in office workers. Eur Spine J. 2014 Apr;23(4):786-93. doi: 10.1007/s00586-014-3212-3. Epub 2014 Feb 4. PMID 24492949
- [Background] Healy GN, Dunstan DW, Salmon J, Cerin E, Shaw JE, Zimmet PZ, Owen N. Breaks in sedentary time: beneficial associations with metabolic risk. Diabetes Care. 2008 Apr;31(4):661-6. doi: 10.2337/dc07-2046. Epub 2008 Feb 5. PMID 18252901
- [Background] Bongers PM, de Winter CR, Kompier MA, Hildebrandt VH. Psychosocial factors at work and musculoskeletal disease. Scand J Work Environ Health. 1993 Oct;19(5):297-312. doi: 10.5271/sjweh.1470. PMID 8296178
- [Background] Hush JM, Michaleff Z, Maher CG, Refshauge K. Individual, physical and psychological risk factors for neck pain in Australian office workers: a 1-year longitudinal study. Eur Spine J. 2009 Oct;18(10):1532-40. doi: 10.1007/s00586-009-1011-z. Epub 2009 Apr 28. PMID 19399537
- [Background] Cagnie B, Danneels L, Van Tiggelen D, De Loose V, Cambier D. Individual and work related risk factors for neck pain among office workers: a cross sectional study. Eur Spine J. 2007 May;16(5):679-86. doi: 10.1007/s00586-006-0269-7. Epub 2006 Dec 8. PMID 17160393
- [Background] Punnett L, Pruss-Utun A, Nelson DI, Fingerhut MA, Leigh J, Tak S, Phillips S. Estimating the global burden of low back pain attributable to combined occupational exposures. Am J Ind Med. 2005 Dec;48(6):459-69. doi: 10.1002/ajim.20232. PMID 16299708
- [Background] Buckle P. Ergonomics and musculoskeletal disorders: overview. Occup Med (Lond). 2005 May;55(3):164-7. doi: 10.1093/occmed/kqi081. PMID 15857895
- [Background] Maniadakis N, Gray A. The economic burden of back pain in the UK. Pain. 2000 Jan;84(1):95-103. doi: 10.1016/S0304-3959(99)00187-6. PMID 10601677
- [Background] Samad NIA AH, Moin S, Tamrin SBM and Hashim Z. Prevalence of Low Back Pain and its Risk Factors among School Teachers. American Journal of Applied Sciences. 2010;7(5):634-
- See also: Raosoft, Inc. (2004). Sample size calculator. — http://www.raosoft.com/samplesize.html